CLINICAL TRIAL: NCT00903656
Title: Lapatinib Plus Caelyx in Patients With Advanced Metastatic Breast Cancer Following Failure of Trastuzumab Therapy - a Phase II Study
Brief Title: Lapatinib Plus Caelyx in Patients With Advanced Metastatic Breast Cancer Following Failure of Trastuzumab Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Caelyx was not available anymore
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MBC-5; EudraCT 2008-004530-25
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2013-12-24 (Estimated); Status verified 2013-12

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; Her2; Lapatinib; Caelyx; cardiotoxic
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caelyx/Lapatinib (Experimental)
  Interventions: Drug: doxorubicinhydrochloride, Lapatinib

INTERVENTIONS:
Drug: doxorubicinhydrochloride, Lapatinib — Lapatinib 1250mg/d p.o. Caelyx 40 mg/m² i.v. q4w for a maximum of 6 cycles

SUMMARY:
The aim of this study is to evaluate the potential of a Lapatinib plus Caelyx combination therapy as an effective and safe therapeutic regimen with a favourable cardiotoxicity profile, in the treatment of metastatic breast cancer following failure of prior trastuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, age ≥ 18 years
* Advanced or metastatic breast cancer, histologically confirmed
* Documented HER2 overexpression (IHC 3+ and/or FISH positive)
* At least one measurable lesion according to RECIST criteria. Patients with bone-only lesions are not eligible for study entry
* Documented disease progression
* Patients may have no more than 1 line of palliative treatment, however prior therapies must include trastuzumab in adjuvant or metastatic setting
* Life expectancy of at least 12 weeks
* Performance status 0-1
* Cardiac ejection fraction >= 50% as measured by echocardiogram or MUGA scan
* Adequate hematology, liver and renal function

Exclusion Criteria:

* Pregnant or lactating women
* Serious medical or psychiatric disorders that would interfere with the patient's safety or informed consent
* Severe cardiac disease (uncontrolled angina, arrhythmia, chronic heart failure (CHF) or cardiac disease requiring a device)
* Ejection fraction below the institutional normal limit
* Maximum cumulative dose of 360 mg/m2 for doxorubicin and 720 mg/m2 for epirubicin
* Active bacterial, viral or fungal infection
* Patients with clinically apparent brain metastases
* Positivity for HIV, Hepatitis B or C
* History of other malignancy; patients who have been disease-free for 5 years
* Concurrent cancer therapy (chemotherapy, radiation therapy, immunotherapy, biologic therapy) or concurrent treatment with an investigational drug or participation in another clinical trial
* Known hypersensitivity to the study drugs Lapatinib and Caelyx or their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Efficacy of a Lapatinib plus Caelyx combination regimen in the treatment of advanced metastatic breast cancer, in terms of overall response rates (complete or partial response)determined by RECIST

SECONDARY OUTCOMES:
Safety profile
Occurrence of clinically apparent brain metastases
Overall survival, progression free survival, clinical benefit (CR, PR or stable disease for at least 24 weeks)
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Alois Lang, Dr, Principal Investigator — LKH Feldkirch; Rainhard Ziebermayr, Dr., Principal Investigator — KH Elisabethinen Linz; Richard Greil, Prof., Principal Investigator — Uniklinik Salzburg; Hellmut Samonigg, Prof., Principal Investigator — Univ. Klinikum Graz; Michael Fridrik, Doz., Principal Investigator — AKH Linz
Locations (1):
- Uniklinik Salzburg, Salzburg, Salzburg, Austria